CLINICAL TRIAL: NCT04430933
Title: A Phase 1/2 Study of NC318 in Combination With Chemotherapy for Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Safety and Tolerability Study of NC318 in Combination With Chemotherapy for Subjects With Advanced or Metastatic NSCLC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Upon reviewing current available combo studies, the sponsor decided to prioritize different combo study.
Sponsor: NextCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC318-02
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Advanced or Metastatic Solid Tumors; Non-Small Cell Lung Cancer
Keywords: Advanced Cancer; NC318; Metastatic Cancer; Non-Small Cell Lung Cancer; NSCLC; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Pemetrexed; Carboplatin; Taxes; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NC318 + Pemetrexed/Carboplatin (Experimental): NC318 at various dose strengths administered on the first day of each 21 day cycle in combination with pemetrexed/carboplatin
  Interventions: Drug: NC318; Drug: Pemetrexed/Carboplatin
- NC318 + Nab-paclitaxel/carboplatin (Experimental): NC318 at various dose strengths administered on the first day of each 21 day cycle in combination with Nab-paclitaxel/carboplatin
  Interventions: Drug: NC318; Drug: Nab paclitaxel/Carboplatin
- NC318 + Docetaxel (Experimental): NC318 at various dose strengths administered on the first day of each 21 day cycle in combination with Docetaxel
  Interventions: Drug: NC318; Drug: Docetaxel

INTERVENTIONS:
Drug: NC318 — NC318 is an experimental antibody drug that will be administered by IV infusion on the first day of each 21 day cycle
Drug: Pemetrexed/Carboplatin — Pemetrexed/Carboplatin will be administered per the approved respective product label following the infusion of NC318 on the first day of each 21 day cycle
  Arms: NC318 + Pemetrexed/Carboplatin
Drug: Nab paclitaxel/Carboplatin — Nab-paclitaxel/Carboplatin will be administered per the approved respective product label following the infusion of NC318 on the first day of each 21 day cycle
  Arms: NC318 + Nab-paclitaxel/carboplatin
Drug: Docetaxel — Docetaxel will be administered per the approved product label following the infusion of NC318 on the first day of each 21 day cycle
  Arms: NC318 + Docetaxel

SUMMARY:
This research study is studying an investigational drug, NC318, as a possible treatment for subjects with advanced or metastatic non-small cell lung cancer in combination with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older.
* Willingness to provide written informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Have a life expectancy of at least 6 months
* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Disease progression after receipt of a prior systemic immunotherapy such as monoclonal antibodies targeting PD-1, PD-L1, CTLA-4 or other immune modulators with or without chemotherapy.
* Presence of measurable disease based on RECIST v1.1. Tumor lesions - situated in a previously irradiated area, or in an area subjected to other locoregional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* After dose escalation, subject must be willing to undergo pretreatment and on-treatment tumor biopsies (core or excisional). Note: A baseline biopsy obtained for other purposes (i.e., not an NC318-02 study procedure) before signing consent may be utilized if the subject has not had any intervening systemic therapy from the time of the biopsy to the start of treatment with the medical monitor's approval.
* Female subjects of childbearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as ≥ 12 months of amenorrhea) must have a negative serum pregnancy test at screening. All female and male subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy or fathering children (with at least 99% certainty) from screening through 60 days after the last dose of study drug.

Exclusion Criteria:

* Inability to comprehend or unwilling to sign the Informed Consent Form.
* Received more than 1 prior line of systemic anti-cancer therapy for Stage IIIB/IIIc/IV or recurrent NSCLC disease (does not include adjuvant or neoadjuvant treatments).
* Requires concurrent radiation or other anticancer therapy
* Screening laboratory values of:

  1. Absolute neutrophil count < 1.5 × 10^9/L
  2. Platelets < 100 × 10^9/L
  3. Hemoglobin < 9 g/dL or < 5.6 mmol/L
  4. Serum creatinine > 1.5 × institutional upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 × ULN
  6. Total bilirubin ≥ 1.5 × ULN unless conjugated bilirubin ≤ ULN (conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN). If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin.
  7. International normalized ratio (INR) or prothrombin time (PT) > 1.5 × ULN
  8. Activated partial thromboplastin time (aPTT) > 1.5 × ULN
* Transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days before the first administration of study drug.
* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

  * ≤ 21 days for chemotherapy or radiation therapy. Subjects must also not require chronic use of corticosteroids and must not have had radiation pneumonitis because of a treatment. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with medical monitor approval. Note: Bisphosphonates and denosumab are permitted medications.
  * ≤ 7 days for immune-suppressive-based treatment for any reason. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted. Note: The use of physiologic corticosteroid replacement therapy may be approved after consultation with the medical monitor.
  * ≤ 28 days or 5 half-lives (whichever is longer) for prior ICI.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting therapy. Note: Subjects with stable chronic conditions (≤ Grade 2) not expected to resolve (such as neuropathy and alopecia) are exceptions and may enroll. Note: Subjects with a history of any grade immune-related ocular AE (e.g., episcleritis, scleritis, uveitis) will be excluded. Note: Subjects with a history of a Grade 3 or higher immune-related AE from prior immunotherapies are excluded.
* History of recurrent Grade 2 pneumonitis attributed to prior treatment with immune checkpoint inhibitor therapy
* Receipt of a live vaccine within 30 days of planned start of study therapy. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Active autoimmune disease that required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Subjects who have not required systemic treatment in the past 2 years may be eligible with approval of the medical monitor. Note: Subjects with hyper/ hypothyroidism are eligible to participate. Note: Replacement and symptomatic therapies (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic immune suppressive therapy and are allowed.
* Known active CNS metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days before the first dose of study drug and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases or CNS edema, and have not required steroids for at least 7 days before the first dose of study drug.
* Known concurrent malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry apart from cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the subject has been disease-free for > 1 year, after treatment with curative intent.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.
* Active infection requiring systemic therapy.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation. HBV-DNA and HCV-RNA must be undetectable. Subjects cannot be positive for HBV-DNA, HCV-RNA, hepatitis B surface antigen, or anti-hepatitis B core antibody. Note: Subjects with no prior history of hepatitis B infection who have been vaccinated against hepatitis B and who have a positive antibody against hepatitis B surface antigen test as the only evidence of prior exposure may participate in the study.
* Known history of HIV (HIV 1 or HIV 2 antibodies).
* Known allergy or reaction to any component of study drug or formulation components.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 60 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-06 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0 | 14 months
  Frequency, duration, and severity of treatment-emergent adverse events (AEs)

SECONDARY OUTCOMES:
Objective Response Rate per RECIST | 14 months
  Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST (mRECIST) v1.1
Duration of Response per RECIST | 14 months
  Duration of Response (DoR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST (mRECIST) v1.1
Disease Control Rate per RECIST | 14 months
  Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST (mRECIST) v1.1
Progression-Free Survival per RECIST | 14 months
  Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST (mRECIST) v1.1
Overall Survival per RECIST | 14 months
  Overall Survival (OS) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST (mRECIST) v1.1
Maximum Plasma Concentration (Cmax) of NC318 | 14 months
  To evaluate the Maximum Plasma Concentration (Cmax) of NC410

CONTACTS AND LOCATIONS:
Overall Officials: Sol Langermann, PhD, Study Director — NextCure, Inc.

IPD SHARING:
Plan to Share IPD: No